CLINICAL TRIAL: NCT01671878
Title: Characterization of the Postprandial Glucose and Insulin Responses to Test Foods in Lean and Overweight Subjects
Brief Title: Glucose and Insulin Responses to Test Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GIl1244
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Glucose Response; Insulin Response
MeSH Terms: interventions — Edible Grain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference Glucose (Other): Glucose standard
  Interventions: Other: Reference Glucose
- Test Food 1 (Experimental): Cereal
  Interventions: Other: Test Food 1 (Cereal)
- Test Food 2 (Experimental): Biscuit
  Interventions: Other: Test Food 2 (Biscuit)

INTERVENTIONS:
Other: Reference Glucose
  Arms: Reference Glucose
Other: Test Food 1 (Cereal)
  Arms: Test Food 1
Other: Test Food 2 (Biscuit)
  Arms: Test Food 2

SUMMARY:
In this study, postprandial glucose and insulin responses of different foods will be measured in individuals with varying body weight.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be non-smoking males or non-pregnant females aged 20-45y, with normal glycemia and in good health. A total of 12 participants will be included, where approximately half will be male & half female, and half normal weight (BMI > 19.0 and < 25.0) and half overweight but not obese (BMI > 25.0 and < 30). Thus, no fewer than 5 male, 5 female, 5 normal weight and 5 overweight but not obese subjects will be included. Additional inclusion criteria will include:
* Absence of diabetes, impaired glucose tolerance and impaired fasting glucose, defined as having a fasting plasma glucose < 5.6 mmol/L (100 mg/dL) AND plasma glucose levels < 7.8 mmol/L (140 mg/dL) 2h after consumption of a 50 g glucose drink (OGTT will be administered during the screening visit)
* Systolic blood pressure 100-150 mmHg inclusive
* Diastolic blood pressure 60-90 mmHg inclusive
* Resting heart rate 50-90 beats/min inclusive after 3 minute rest
* Able to refrain from eating legumes and drinking alcohol the day before each test session
* Fasting triglycerides < 2.0 mmol/L (178 mg/dL)
* Fasting HDL cholesterol > 0.9 mmol/L (35 mg/dL) for males and > 1.1mmol/L (42 mg/dL) for females
* Fasting LDL cholesterol < 5.0 mmol/L (193 mg/dL)
* AST and ALT < 120% of upper limit of normal (ULN)
* hsCRP < 10 mg/L
* Urea and creatinine < 150% ULN

Exclusion Criteria:

* failure to meet any one of the inclusion criteria
* age less than 18 or over 45 years
* known history or AIDS, hepatitis, diabetes or a heart condition
* participants using medications or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results
* participants who cannot or will not comply with the experimental procedures or do not follow GI Labs safety guidelines.
* Food allergies of any kind
* General anaesthesia in the month prior to inclusion.
* Smokers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Postprandial Glucose Response | 3 hours

SECONDARY OUTCOMES:
Postprandial Insulin Response | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada